CLINICAL TRIAL: NCT02328053
Title: Clinical & Visual Outcomes of Collagen Cross Linking for Fungal Keratitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aravind Eye Care System (Other)
Responsible Party: Principal Investigator, Dr.N.Venkatesh Prajna, Chief Cornea Services, Aravind Eye Care System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2013019CLI
Record Dates: First submitted 2014-12-13; First posted 2014-12-31 (Estimated); Last update posted 2014-12-31 (Estimated); Status verified 2014-12

CONDITIONS: Mycotic Corneal Ulcer
Keywords: fungal keratitis; collagen cross linking
MeSH Terms: interventions — Natamycin; Voriconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagen crosslinking group (Experimental): patients not resolving to standard antifungal therapy were assigned to receive adjuvant collagen crosslinking with riboflavin and Ultraviolet-A along with topical medical therapy
  Interventions: Procedure: collagen crosslinking group; Drug: Topical anti-fungal therapy
- standard medical therapy (Active Comparator): patients were continued on topical antifungal therapy namely Natamycin eye drops and voriconazole eye drops
  Interventions: Drug: Topical anti-fungal therapy

INTERVENTIONS:
Procedure: collagen crosslinking group — collagen crosslinking with riboflavin and Ultraviolet A
  Other Names: CXL, C3R
  Arms: Collagen crosslinking group
Drug: Topical anti-fungal therapy — topical antifungal medications like natamycin eye drops and voriconazole eye drops
  Other Names: natamycin, voriconazole

SUMMARY:
The study is a randomised control trial to assess the visual and clinical outcomes of collagen cross linking in fungal keratitis. Fungal keratitis is a major cause of corneal blindness in India and the therapeutic options available are minimal to handle the advanced complications and sequalae caused by the disease.The antimicrobial and tissue remodeling role of corneal cross linking was demonstrated by several studies earlier,we anted to specifically assess the role of corneal cross linking in non resolving fungal keratitis in prevention of perforation and enhancement of healing process.

DETAILED DESCRIPTION:
Patients with culture positive deep stromal fungal keratitis not responding to appropriate medical therapy for a period of two weeks were randomized to receive or not receive adjuvant CXL. The medical therapy was continued in both the groups and were followed up for 6 weeks after randomization. Healing of the ulcer was taken as successful outcome, while perforation and increase in ulcer size of more than 2 sq.mm from the baseline was considered as treatment failure.

ELIGIBILITY:
Inclusion Criteria:

* Ulcer size more than 5 mm
* Ulcer depth upto 70% of stromal depth
* Corneal thickness of 400 microns and above

Exclusion Criteria:

* Corneal thickness of below 400 microns
* Ulcers involving the limbus
* Pregnant women
* Children below the age of 18 years

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-02; Primary Completion 2015-07 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
size of infiltrate or scar, corneal structural integrity | 6 months

SECONDARY OUTCOMES:
visual acuity | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Venkatesh Prajna, DNB,FRCS, Principal Investigator — CHIEF CORNEA SERVICES
Locations (1):
- Aravind Eye Hospital, Madurai, Tamil Nadu, India

REFERENCES:
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558
- [Derived] Uddaraju M, Mascarenhas J, Das MR, Radhakrishnan N, Keenan JD, Prajna L, Prajna VN. Corneal Cross-linking as an Adjuvant Therapy in the Management of Recalcitrant Deep Stromal Fungal Keratitis: A Randomized Trial. Am J Ophthalmol. 2015 Jul;160(1):131-4.e5. doi: 10.1016/j.ajo.2015.03.024. Epub 2015 Apr 1. PMID 25841317